CLINICAL TRIAL: NCT00322959
Title: Effect of Tai-Chi-Chuan on Differentiation and Maturation of Human Dendritic Cells
Brief Title: Tai-Chi-Chuan on Differentiation and Maturation of Dendritic Cells
Status: Completed | Type: Observational
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Yu-Jen Chen, Mackay Memorial Hospital
Other Study IDs: MMH-I-S-056
Record Dates: First submitted 2006-05-05; First posted 2006-05-08 (Estimated); Last update posted 2008-09-22 (Estimated); Status verified 2008-09

CONDITIONS: Immunity
Keywords: dendritic cells; Tai-Chi-Chuan

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Tai-Chi-Chuan (TCC), a branch of traditional Chinese martial arts, has been widely practiced since the 17th century. Recent studies have shown that TCC can improve cardiorespiratory function, muscle strength, humoral and cellular immunity, metabolic response and mental control.

Cultured monocytes from blood or bone marrow can be triggered to differentiate to myeloid dendritic cells (DC). DCs are specialized leukocytes for presenting antigens to quiescent, naive, and memory T cells, and they play pivotal roles in the induction of cell-mediated as well as humoral immune responses in vivo. Mature DCs have a capacity for initiating immunity or tolerance, which depends on their activation state.

In this study we will investigate the effect of TCC on DC differentiation in the peripheral blood obtained from the healthy donors who take part with and without TCC exercise. The distribution of various DC sub-populations (myeloid DC and plasmacytoid cell) will be analyzed by detecting surface marker expression.

DETAILED DESCRIPTION:
Introduction

Tai-Chi-Chuan (TCC), a branch of traditional Chinese martial arts, has been widely practiced since the 17th century. TCC gradually evolved into many styles, the Chen style is the oldest and the Yang style is the most popular. The practice of TCC was originally related to concerns about physical fitness and the capacity for self defense. Over the centuries, it has become far more focused on the homoeostasis of the body's internal environment. The interaction between mind and body has long been seen as more important than the development of any martial arts skills. Classical TCC consists of many complex postures, and performing a complete set takes 20 to 30 minutes. A simplified form of TCC was developed to facilitate promotion in 1956 (1), however, simplified TCC have lesser training benefits owing to reduction of exercise intensity and duration. TCC has been considered as a practice of medico-athletics, which can improvement of physical condition and treatment of certain chronic diseases. Exercise has definite effects on the health of human, but appropriate forms are scarce. Recent studies have shown that TCC can improve cardiorespiratory function (2-4), muscle strength (5), humoral and cellular immunity (6-8), metabolic response (9), and mental control (10). Studies used TCC postures for training showed that the exercise intensity of TCC training is moderate (2). A well designed study for TCC on human health, especially whether TCC improve immune response or not, will be processed in this project.

Dendritic cells (DCs) are specialized leukocytes for presenting antigens to quiescent, naive, and memory T cells, and they play pivotal roles in the induction of cell-mediated as well as humoral immune responses in vivo (11). The exceptional ability of DCs to stimulate T cells in vitro and in vivo is attributed, at least in part, to their ability to capture antigen, to migrate into lymphoid organs, and to express high levels of immunostimulatory molecules, such as major histocompatibility complex (MHC) class II, B7-1, B7-2, and IL-12 (11,12). Immature DCs, such as Langerhans cells of the skin, capture and process antigens very efficiently (13). Upon exposure to various microbial and inflammatory products (eg, lipopolysaccharide [LPS], IL-1, TNF-alpha), DCs mature and migrate into lymphoid tissues to interact with T and B cells (14-17).

In this study we will investigate the effect of Tai-Chi-Chuan (TCC) on DC differentiation in the peripheral blood obtained from the healthy donor who take part with and without TCC exercise. Subjects who practice with or without Yang TCC will be assessed their distribution of various DC sub-populations (myeloid DC and plasmacytoid cell) and their activation state will be analyzed by detecting surface marker expression.

The potential of this study is to demonstrate the immunomodulatory activity of TCC, a novel sport in Chinese for thousand years.

Materials and methods

1. Subjects and study design. Yang TCC practitioner who keep practicing at least 3 times a week for more than 3 years will be recruited.
2. Cardiopulmonary fitness measurement during TCC practice. To determine the exercise intensity and cardiopulmonary fitness of the classical form of Yang TCC, HP responses and VO2max will be measured during TCC exercise. Lactate response before and immediately after TCC practice will be measured. The Cosmed K4 system (Cosmed s.r.l., Rome, Italy) consists of a photoelectric turbine flowmeter will be used to calculate the minute ventilation, and measure the number of expiratory cycles per minute. Cardiorespiratory parameters including heart rate, minute ventilation (VE), oxygen uptake, carbon dioxide production (VCO2), will be also measured.
3. Cell preparation. The mononuclaer cells of blood will be isolated by using centrifugation on a density gradient (Ficoll-Hypaque, 1.077 gm/ml, Pharmacia Fine Chemicals). DCs will be isolated by using CD11c-conjugated MACS magnetic beads.
4. Assess the distribution of various DC sub-populations. Myeloid DC (CD11c+) and plasmacytoid cells (CD123+), which are excluded by lineage markers (CD3，CD14，CD16，CD19，CD20，CD56) will be analyzed by detecting surface marker expression with flow cytometer.

References:

1. China Sports. Simplified "Taijiquan". 1983:1-5. Bejing, China Publications Center.
2. Lan C, Chen SY, Lai JS, Wong MK. Heart rate responses and oxygen consumption during Tai Chi Chuan practice. Am J Chin Med 2001;29:403.
3. Lai JS, Lan C, Wong MK, Teng SH. Two-year trends in cardiorespiratory function among older Tai Chi Chuan practitioners and sedentary subjects. J Am Geriatr Soc 1995;43:1222.
4. Gong L, Qian J, Zhang J, et al. Changes in heart rate and electrocardiogram during Taijiquan exercise. Chin Med J 1981;94:589.
5. Wolfson L, Whipple R, Derby C, et al. Balance and strength training in older adults: intervention gains and Tai Chi maintenance. J Am Geriatr Soc 1996;44:498.
6. Sun X, Xu Y, Zhu R. Detection of ZC resette-forming lymphocytes in the healthy aged with TaichiQuan (88 style) exercise. J Sports Med Physic Fit 1990;30:401.
7. Zhang GD. The impacts of 48-form Tai Chi Chuan and Yi Qi Yang Fei Gong on the serum levels of IgG, IgM, IgA and Ig E in human. Journal of Beijing Institute of Physical Education 1990;4:12.
8. Sun X, Xu Y, Xia Y. Determination of E-resette-forming lymphocytes in aged subjects with Taichiquan exercise. Int J Sports Med 1989;10:217.
9. Zhou D, Shephard RJ, Plyley MJ, et al. Cardiorespiratory and metabolic responses during Tai Chi Chuan exercise. Can J Appl Sport Sci 1984;9:7.
10. Xu S, Fan Z. Physiological studies of Tai Ji Quan in Cina. In: Qu M, Yu C, eds. China's sports medicine. Basel, New York: Karger 1988:70.
11. Banchereau J, Steinman RM. Dendritic cells and the control of immunity. Nature 1998;392:245.
12. Hart DN. Dendritic cells: unique leukocyte populations which control the primary immune response. Blood 1997;90:3245.
13. Albert ML, Pearce SF, Francisco LM, et al. Immature dendritic cells phagocytose apoptotic cells via avb5 and CD36, and cross-present antigens to cytotoxic T lymphocytes. J Exp Med 1998;188:1359.
14. Jonuleit H, Kuhn U, Muller G, et al. Pro-inflammatory cytokines and prostaglandins induce maturation of potent immunostimulatory dendritic cells under fetal calf serum-free conditions. Eur J Immunol. 1997;27:3135.
15. Kato T, Yamane H, Nariuchi H. Differential effects of LPS and CD40 ligand stimulations on the induction of IL-12 production by dendritic cells and macrophages. Cell Immunol 1997;181:59.
16. Cella M, Scheidegger D, Palmer-Lehmann K, Lane P, Lanzavecchia A, Alber G. Ligation of CD40 on dendritic cells triggers production of high levels of interleukin-12 and enhances T cell stimulatory capacity: T-T help via APC activation. J Exp Med 1996;184:747.
17. Labeur MS, Roters B, Pers B, et al. Generation of tumor immunity by bone marrow-derived dendritic cells correlates with dendritic cell maturation stage. J Immunol 1999;162:168.

ELIGIBILITY:
Inclusion Criteria:

* Yang TCC practitioner who keep practicing at least 3 times a week for more than 3 years
* Healthy subjects as controls

Exclusion Criteria:

* Who have a history of significant cardiovascular, pulmonary, and musculoskeletal diseases

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: TCC practitioner and Healthy subjects as controls
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2004-08; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Jen Chen, MD, PhD, Principal Investigator — Mackay Memorial Hospital
Locations (1):
- Department of Medical Research, Mackay Memorial Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Lee JJ, Liao HF, Yang YC, Liu CL, Chen YY, Lin CP, Chen YJ. Platonin modulates differentiation and maturation of human monocyte-derived dendritic cells. Int Immunopharmacol. 2006 Feb;6(2):287-93. doi: 10.1016/j.intimp.2005.08.016. Epub 2005 Sep 15. PMID 16399634